CLINICAL TRIAL: NCT01779310
Title: Clinical Pathway for Alzheimer's Disease in China (CPAD): A 8-week Multi-center Registry Study to Investigate AD Diagnostic Pattern in Chinese Local Real Clinical Practice
Brief Title: Clinical Pathway for Alzheimer's Disease in China (CPAD)
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Beijing Novartis Pharma (Industry)
Responsible Party: Principal Investigator, Huali Wang, Associate Professor, Peking University
Other Study IDs: CENA731DCN01T
Record Dates: First submitted 2013-01-24; First posted 2013-01-30 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alzheimer's disease: Outpatients with clinically significant cognitive impairment per judgment of the participating physicians are enrolled.

SUMMARY:
There are guidelines on the management of AD in China, the evidence adopted in the guidelines are mostly from the trials conducted in other countries due to very limited Chinese data available for local systematic review. Therefore, more local evidence on dementia care is needed for the development of an evidence-based guideline appropriate for people living in China. Meanwhile, the inadequate implementation of the current AD guideline, which results in the low diagnostic rate and high diagnostic leakage, may bring about extra barriers for AD patients to access dementia care service in different areas nationwide. However, there is no data on the clinical pathway about how physicians follow the dementia guideline in the routine practice.

Therefore, research is needed to learn clinical diagnostic process and treatment patterns of physicians to people with AD in routine practice and help address the low accurate rate of AD clinical diagnosis and low anti-dementia drug prescription in the real world and support guideline development.

DETAILED DESCRIPTION:
Outpatients who are visiting memory clinics and who are judged by physicians with clinically significant cognitive impairment will be invited to join the study during the study recruiting period (with informed consent signed).

* Patients enrolled into the study will be evaluated and diagnosed by participating physicians and may or may not be prescribed with therapy (pharmaceutical and/or non-pharmaceutical) based on physicians' medical judgment.
* For patients with routine clinical follow-up visits, their medical charts will be reviewed for documentation. The procedures of making diagnosis and developing treatment scheme will be retrieved and documented in clinical report form (CRF). Additional procedures ordered by the participating physician at current visits will also be documented in CRF.

All participants will be followed twice after baseline visit to re-evaluate and confirm the initial diagnosis (where applicable), and to record compliance to treatment scheme, including the process of medication titration.

This study does not recommend nor restrict any specific treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients with clinically significant cognitive impairment per independent judgment of participating physicians;
* Aged 45 year old and above;
* Willing to receive 2 follow-up visits;
* Having at least one informant or caregiver accompanying during each visit;
* Willing to join the study and sign the informed consent prior to the study.

Exclusion Criteria:

* Cognitive impairment is likely or identified as secondary to other disease condition(s) than AD (including but not limited to stroke, Parkinson's disease, brain trauma, central nervous system infection, etc.)
* Unwilling to participate in the study;
* Participating other studies during the registry study period.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with clinically significant cognitive impairment per judgment of the participating physicians are registered.
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rate of cognitive assessment administration | 2 months
  rate of cognitive assessment administration for diagnosing dementia

SECONDARY OUTCOMES:
Rate of anti-dementia prescription | 2 months
  rate of anti-dementia prescription for people with dementia

OTHER OUTCOMES:
compliance rate of anti-dementia prescription | 2 months
  rate of continuous using anti-dementia drugs among patients with dementia

CONTACTS AND LOCATIONS:
Overall Officials: Huali Wang, MD/PhD, Principal Investigator — Peking University Institute of Mental Health (Sixth Hospital)
Locations (28):
- China (28):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Mecial College, Huazhong University of Science and Technology, Wuhan, Hebei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Mental Health Center, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Mental Health Center, West China Hospital, Sichuan University, Chengdu, Sichuan
  - General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Ningbo Kangning Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital, Wenzhou Medical College, Wenzhou, Zhejiang